CLINICAL TRIAL: NCT01679496
Title: Fat Quality on Blood Lipids and Immune Response
Acronym: NoMa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo Metropolitan University (Other); Mills DA (Industry)
Responsible Party: Principal Investigator, Stine Marie Ulven, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: REK 2011/1951
Record Dates: First submitted 2012-08-24; First posted 2012-09-06 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Dietary Prevention
Keywords: LDL-cholesterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Food items (Experimental): Food items low in saturated fat and high in polyunsaturated fat
  Interventions: Other: Food items
- Control food items (Placebo Comparator): Food items containing saturated fat and polyunsaturated fat according to a traditional Norwegian diet
  Interventions: Other: Food items

INTERVENTIONS:
Other: Food items — Food items with different fatty acid composition

SUMMARY:
The purpose of this study is to investigate blood LDL-cholesterol and level of inflammatory markers after intake of food items with different fatty acid composition.

ELIGIBILITY:
Inclusion Criteria:

* hsCRP < 10 mg/L
* total cholesterol 5-7.8 mmol/l(50-70 y)
* total cholesterol 5.0-6.9 mmol/l (30-49 y)
* total cholesterol 5.0-6.1 mmol/l (25-29 y)
* LDL-cholesterol at or above 3.5 mmol/l
* triglycerides at or lower 2.6 mmol/l
* BMI 20-35
* Stable bodyweight last 3 months.

Exclusion Criteria:

* Chronic diseases
* fasting glucose > 6.0 mmol/l
* increased ASAT and ALAT
* medications affecting lipidmetabolism and inflammation

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in LDL-cholesterol | Change from baseline after 8 weeks
  Change in LDL-cholesterol when compared to control diet
Change in total cholesterol | Change from baseline after 8 weeks
  Change in total cholesterol when compared to control diet

SECONDARY OUTCOMES:
Inflammatory markers in circulation and at gene expression level in PBMC | Inflammatory markers are measured at baseline and after 8 weeks intervention in circulation and at gene expression level in PBMC
Markers of lipid metabolism at gene expression level in PBMC | Markers of lipid metabolism at gene expression level in PBMC is measured at baseline and after 8 weeks of intervention
Appetite hormones | Appetite hormones is measured at baseline and after 8 weeks of intervention
Gut peptides | Gut peptides are measured at baseline and after 8 weeks of intervention
Metabolites | Metabolites are measured at baseline and after 8 weeks of intervention
  Targeted and untargeted metabolomics will be measured
Whole genome gene expression | whole genome gene expression profiles are measured at baseline and after 8 weeks of intervention
  Microarray

CONTACTS AND LOCATIONS:
Overall Officials: Stine Ulven, PhD, Principal Investigator — University of Oslo; Kirsten B Holven, PhD, Principal Investigator — Department of Nutrition, Institute for Basic Medical Sciences, University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway

REFERENCES:
- [Derived] Pigsborg K, Gurdeniz G, Rangel-Huerta OD, Holven KB, Dragsted LO, Ulven SM. Effects of changing from a diet with saturated fat to a diet with n-6 polyunsaturated fat on the serum metabolome in relation to cardiovascular disease risk factors. Eur J Nutr. 2022 Jun;61(4):2079-2089. doi: 10.1007/s00394-021-02796-6. Epub 2022 Jan 9. PMID 34999928
- [Derived] Ulven SM, Christensen JJ, Nygard O, Svardal A, Leder L, Ottestad I, Lysne V, Laupsa-Borge J, Ueland PM, Midttun O, Meyer K, McCann A, Andersen LF, Holven KB. Using metabolic profiling and gene expression analyses to explore molecular effects of replacing saturated fat with polyunsaturated fat-a randomized controlled dietary intervention study. Am J Clin Nutr. 2019 May 1;109(5):1239-1250. doi: 10.1093/ajcn/nqy356. PMID 31051508